CLINICAL TRIAL: NCT04044053
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE-DOSE, 4-PERIOD, 4-SEQUENCE, CROSSOVER STUDY TO EVALUATE THE RELATIVE BIOAVAILABILITY OF A MODIFIED-RELEASE FORMULATION OF PF-06865571 RELATIVE TO AN IMMEDIATE-RELEASE FORMULATION UNDER FED CONDITIONS, AND TO EVALUATE THE EFFECT OF FASTING ON THE PHARMACOKINETICS OF THE MODIFIED-RELEASE FORMULATION, IN HEALTHY WESTERN AND JAPANESE PARTICIPANTS
Brief Title: Relative Bioavailability Study of a Modified-Release Formulation of PF-06865571 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C2541012; 2019-001426-96 (EudraCT Number)
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Healthy Participants
Keywords: PF-06865571; Relative bioavailability; Modified release; Diacylglycerol acyltransferase; DGAT2; Japanese
MeSH Terms: interventions — ervogastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Relative Bioavailability (Experimental): Each participant will receive 400 mg IR, 400 mg MR, and 50 mg MR in the fed state, and 400 mg MR in the fasted state
  Interventions: Drug: PF-06865571 400 mg Immediate Release (IR) in Fed State; Drug: PF-06865571 50 mg Modified Release (MR) in Fed State; Drug: PF-06865571 400 mg MR in Fed State; Drug: PF-06865571 400 mg MR in Fasted State
- Fasted State (Experimental): Comparison of 400 mg MR in fed and fasted states
  Interventions: Drug: PF-06865571 400 mg MR in Fed State; Drug: PF-06865571 400 mg MR in Fasted State

INTERVENTIONS:
Drug: PF-06865571 400 mg Immediate Release (IR) in Fed State — 400 mg IR dose in fed state
  Arms: Relative Bioavailability
Drug: PF-06865571 50 mg Modified Release (MR) in Fed State — 50 mg MR in fed state
  Arms: Relative Bioavailability
Drug: PF-06865571 400 mg MR in Fed State — 400 mg MR in fed state
Drug: PF-06865571 400 mg MR in Fasted State — 400 mg MR in fasted state

SUMMARY:
This study is an open-label, randomized, single-dose, 4-period, 4-sequence, crossover study in a single cohort of approximately 12 healthy adult participants. The purpose of this study is to evaluate the relative bioavailability of a newly developed modified release (MR) tablet formulation of PF-06865571 relative to an immediate release (IR) tablet formulation of PF-06865571 under fed conditions. In addition, this study will also assess the relative bioavailability of the MR formulation under fasted conditions relative to fed conditions, in healthy adult participants. Study results will be used to determine if the new MR formulation may be suitable for use in future clinical studies with PF-06865571. Healthy adult Japanese participants will also be enrolled in this study to support inclusion of Japanese participants in future clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of non-childbearing potential and male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac tests.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Participants enrolling as Japanese must have 4 biological Japanese grandparents who were born in Japan.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product used in this study (whichever is longer).
* Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* Baseline 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline corrected QT (QTc) interval >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias).
* Participants with any of the following abnormalities in clinical laboratory tests at screening: Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≥1.25× upper limit of normal (ULN); Total bilirubin level ≥1.5× ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Single Dose Maximum Observed Plasma Concentration (Cmax) of PF-06865571 in Healthy Participants | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  All study participants
Single Dose Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06865571 in Healthy Participants | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  All study participants
Single Dose Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC(last)] of PF-06865571 in Healthy Participants | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  All study participants
Single Dose Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC(0-∞)] of PF-06865571 in Healthy Participants | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  All study participants

SECONDARY OUTCOMES:
Single Dose Cmax of PF-06865571 in Healthy Japanese Participants | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  Japanese participants only
Single Dose Tmax of PF-06865571 in Healthy Japanese Participants | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  Japanese participants only
Single Dose AUC(last) of PF-06865571 in Healthy Japanese Participants | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  Japanese participants only
Single Dose AUC(0-∞) of PF-06865571 in Healthy Japanese Participants | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  Japanese participants only
Fasted State Single Dose Cmax of Modified-Release (MR) Formulation of PF-06865571 in Healthy Participants | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  All study participants
Fasted State Single Dose Tmax of MR Formulation of PF-06865571 in Healthy Participants | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  All study participants
Fasted State Single Dose AUC(last) of MR Formulation of PF-06865571 in Healthy Participants | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  All study participants
Single Dose AUC(0-∞) of MR Formulation of PF-06865571 in Healthy Participants | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  All study participants
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline (Day -1) up to 35 days after last dose of study medication
  Treatment-related AEs are any untoward medical occurrences attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Y days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug X was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline (Day -1) and Day 3 of each period
  Laboratory parameters included: hematology (hemoglobin, hematocrit, red blood cell, platelet and white blood cell count, neutrophils, eosinophils, monocytes, basophils and lymphocytes), chemistry (blood urea nitrogen, creatinine, sodium, potassium, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein and serum pregnancy test [for all female participants]) and urine (urine pregnancy test [for all female participants]). Clinical significance of laboratory parameters was determined at the investigator's discretion.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  Vital signs (temperature, respiratory rate, pulse, systolic and diastolic blood pressure) were obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Clinical significance of vital signs was determined at the investigator's discretion.
Number of Participants With Change From Baseline in Electrocardiogram (ECG) Findings | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose
  Criteria for potentially clinically important (PCI) changes in ECG (12-lead) were defined as: no sinus rhythm; PR interval >=220 msec and increase of >=20 msec; QRS interval >=120 msec; QT interval corrected using the Fridericia formula (QTcF) and QT interval corrected using the Bazett's formula (QTcB) >500 msec or increase of >60 msec; heart rate <=45 beats per minute (bpm) or >=120 bpm or decrease/increase of >=15 bpm.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Be-bru, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2541012